CLINICAL TRIAL: NCT01529827
Title: A Phase II Trial of Reduced Intensity Allogeneic Stem Cell Transplantation With Fludarabine, Melphalan and Low Dose Total Body Irradiation
Brief Title: Fludarabine Phosphate, Melphalan, and Low-Dose Total-Body Irradiation Followed by Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 177110; NCI-2011-03563 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Grade III Lymphomatoid Granulomatosis; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Aplastic Anemia; Burkitt Lymphoma; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Grade III Lymphomatoid Granulomatosis; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Congenital Amegakaryocytic Thrombocytopenia; Diamond-Blackfan Anemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Juvenile Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Paroxysmal Nocturnal Hemoglobinuria; Peripheral T-cell Lymphoma; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Secondary Myelofibrosis; Severe Combined Immunodeficiency; Severe Congenital Neutropenia; Shwachman-Diamond Syndrome; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Waldenstrom Macroglobulinemia; Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Anemia, Aplastic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Congenital amegakaryocytic thrombocytopenia; Anemia, Diamond-Blackfan; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Hemoglobinuria, Paroxysmal; Lymphoma, T-Cell, Peripheral; Polycythemia Vera; Primary Myelofibrosis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Severe Combined Immunodeficiency; Neutropenia, Severe Congenital, Autosomal Recessive 3; Shwachman-Diamond Syndrome; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia; Wiskott-Aldrich Syndrome | interventions — fludarabine phosphate; Melphalan; Whole-Body Irradiation; Tacrolimus; Mycophenolic Acid; Methotrexate; merphos; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (reduced intensity allogeneic PBSCT) (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV over 30 minutes on days -5 to -2 and melphalan IV over 30 minutes on day -2. Patients undergo low-dose TBI BID on day -1. TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0. GvHD PROPHYLAXIS: Patients receive tacrolimus IV or PO BID on days -1 to 100 with taper over 4-6 months, MMF PO or IV every 6-8 hours on days -1 to 60, and methotrexate IV over 15 to 30 minutes on days 1, 3, and 6.
  Interventions: Drug: fludarabine phosphate; Drug: melphalan; Radiation: total-body irradiation; Drug: tacrolimus; Drug: mycophenolate mofetil; Drug: methotrexate; Other: laboratory biomarker analysis; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Drug: mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Other: laboratory biomarker analysis — Correlative studies
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSCT
Procedure: peripheral blood stem cell transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
This phase II trial studies how well giving fludarabine phosphate, melphalan, and low-dose total-body irradiation (TBI) followed by donor peripheral blood stem cell transplant (PBSCT) works in treating patients with hematologic malignancies. Giving chemotherapy drugs such as fludarabine phosphate and melphalan, and low-dose TBI before a donor PBSCT helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from the donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cell from a donor can make an immune response against the body's normal cells. Giving tacrolimus, mycophenolate mofetil (MMF), and methotrexate after transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the transplant related mortality (TRM) of this reduced-intensity transplantation (RIT) combination, fludarabine (fludarabine phosphate), melphalan, and TBI in a patient population usually not eligible for a full a myeloablative allogeneic hematopoietic stem cell transplantation (HSCT).

SECONDARY OBJECTIVES:

I. To evaluate clinical response, progression free survival (PFS) at one year, engraftment rate, and graft-versus-host disease (GvHD) incidence with the proposed RIT regimen across a variety of hematological conditions.

II. Correlative studies will include chimerism analysis by molecular analysis and evaluation of immune reconstitution by cytomegalovirus (CMV) dextramer analysis using flow cytometry.

OUTLINE: PREPARATIVE REGIMEN:

Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -5 to -2 and melphalan IV over 30 minutes on day -2. Patients undergo low-dose TBI twice daily (BID) on day -1.

TRANSPLANTATION:

Patients undergo allogeneic PBSCT on day 0.

GvHD PROPHYLAXIS:

Patients receive tacrolimus IV or orally (PO) BID on days -1 to 100 with taper over 4-6 months, MMF PO or IV every 6-8 hours on days -1 to 60, and methotrexate IV over 15-30 minutes on days 1, 3, and 6. After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a histology documented hematologic malignancy or marrow disorder

BONE MARROW FAILURE DISORDERS:

* Acquired bone marrow failure disorders include aplastic anemia, paroxysmal nocturnal hemoglobinuria (PNH) * Primary allogeneic HSCT is appropriate for selected patients with severe aplastic anemia; however, patients with aplastic anemia must have failed at least one cycle of standard immunosuppressive therapy with calcineurin inhibitor plus anti-thymocyte globulin (ATG) if a fully matched donor is available * Patients with PNH should not be eligible for a myeloablative HSCT
* Hereditary bone marrow failure disorders include Diamond-Blackfan Anemia, Shwachman-Diamond Syndrome, Kostmann Syndrome, congenital Amegakaryocytic Thrombocytopenia; Fanconi Anemia or related chromosomal breakage syndrome, Dyskeratosis Congenital are excluded from this study die to their poor deoxyribonucleic acid (DNA) repair capacity * Fanconi anemia or related chromosomal breakage syndrome: positive chromosome breakage analysis using diepoxybutane (DEB) or mitomycin C if applicable * Dyskeratosis Congenita: diagnosis is supported by using either telomerase RNA component (TERC) gene mutation in autosomal dominant Dyskeratosis Congenita or X-linked DKC1 gene mutation
* Other non-malignant hematologic or immunologic disorders that require transplantation * Quantitative or qualitative congenital platelet disorders (including but not limited to congenital amegakaryocytopenia, absent-radii syndrome, Glanzmann's thrombasthenia) * Quantitative or qualitative congenital neutrophil disorders (including but not limited to chronic granulomatous disease, congenital neutropenia) *Congenital primary immunodeficiency syndrome, Wiskott-Aldrich syndrome, CD40 ligand deficiency, T-cell deficiencies)

ACUTE LEUKEMIAS:

* Subjects must be ineligible for or unable to receive a conventional myeloablative transplantation
* Resistant or recurrent disease after at least one standard combination chemotherapy OR first remission patients at high risk of relapse * Acute myeloid leukemia (AML)
* antecedent myelodysplastic syndrome, secondary AML, high risk cytogenetic abnormalities or normal cytogenetics with high-risk molecular mutations (e.g., fms-like tyrosine kinase3-internal tandem duplication [Flt3-ITD] mutation) * Acute lymphocytic leukemia (ALL)
* high or standard risk ALL

CHRONIC MYELOID LEUKEMIA (CML):

* Chronic phase (intolerant or unresponsive to imatinib and/or other tyrosine kinase inhibitors), second chronic phase or accelerated phase who are ineligible for conventional myeloablative transplantation

MYELOPROLIFERATIVE AND MYELODYSPLASTIC SYNDROME (MDS):

* Myelofibrosis (with/without splenectomy) with intermediate to high risk features
* Advanced polycythemia vera nor responding to standard therapy
* MDS with lower International Prognostic Scoring System (IPSS) score of intermediate (Int)-2 or higher
* MDS with lower IPSS score Int-1 or less with severe clinical features such as severe neutropenia or thrombocytopenia or high risk chromosome abnormalities such as monosomy 7
* Secondary MDS with any IPSS scores
* Chronic myelomonocytic leukemia

LYMPHOPROLIFERATIVE DISEASE:

* Chronic lymphocytic leukemia (CLL), low-grade non-Hodgkin lymphoma (NHL) (recurrent or persistent) fludarabine refractory or with less than 6 months duration or complete remission (CR) between courses of conventional therapy
* Multiple myeloma (progressive disease after autologous stem cell transplant, tandem allogeneic transplant after prior autologous stem cell transplant)
* Waldenstrom's macroglobulinemia (failed one standard regimen)
* High grade NHL and diffuse large B-cell lymphoma (DLBCL)
* Not eligible for conventional myeloablative HSCT OR failed autologous HSCT
* First remission lymphoblastic lymphoma, or small, non-cleaved cell lymphoma or mantle cell lymphoma

HODGKIN LYMPHOMA:

* Received and failed front-line therapy
* Failed or were not eligible for autologous transplantation DONOR: Permissible human leukocyte antigen (HLA) matching: related donors
* single antigen mismatch at HLA A, B, or DRB1; unrelated donors
* a single antigen mismatch at HLA A, B, or C, +/- additional single allele level mismatch at A, B, V or DRB1
* Minimum goal for peripheral blood stem cells (PBSC) dose is 2 x 10^6 CD34+ cells/kg of recipient weight; minimum goal for the marrow dose is 1 x 10^8 nucleated cells/kg of recipient weight
* No serious uncontrolled psychiatric illness
* No concomitant active malignancy that would be expected to require chemotherapy within 3 years of transplant (other than non-melanoma skin cancer)
* Non-pregnant and non-nursing woman; (women or men with reproductive potential should agree to use an effective means of birth control)
* Patients who have failed a prior autologous or allogeneic transplant are eligible; however, at least 90 days must have elapsed between the start of this reduced intensity conditioning regimen and the last transplant if patient had a prior autologous or myeloablative allogeneic bone marrow transplant (BMT)
* At least 2 weeks since prior chemotherapy, radiation treatment and/or surgery
* Informed consent

DONOR: Compatibility at the four most informative HLA loci:

A, B, C and DRB1 are important for reducing the risk of GVHD and successful transplant outcomes; the A, B, C and DRB1 loci comprise 8 possible alleles (a haplotype being inherited from each parent); one additional locus, HLA-DQ, is also typed to ascertain haplotypes and assist in the search for a compatible donor; however mismatching at DQ has not been shown to be associated with adverse outcomes; high resolution molecular typing (at the allele level) is now the standard of care for unrelated donor searches and allows greater refinement of the search strategy

DONOR: Matched related donor:

a single antigen mismatch at A, B, or the DR transplant from a family member is associated with a higher risk of GVHD but similar overall survival when compared to full identity at these 3 regions; related donor/recipient pairs must be matched at 5 of 6 HLA antigens (A, B, DRB1)

DONOR: Unrelated Donor:

When evaluating patients for unrelated donor transplant, the higher degree of matching, the lower risk of GvHD; the A, B, C, DRB1 and DQB1 loci, comprising 10 possible antigen (with alleles), will be typed for all unrelated transplants; given the higher risk of TRM in mismatched transplants, RIT is often the best way to mitigate the risk; data from the National Marrow Donor Program makes it possible to estimate the risk of donor-recipient HLA mismatch at the allele or antigen level; the higher risk from HLA-mismatching must be balanced against the clinical urgency and the patient's risk by the transplant team; at this time, antigen level mismatches at DQB1 do not affect outcomes and will not be used for matching purposes for donor selection; thus, the matching required will be at the HLA A, B, C and DRB1 (8 loci); for this protocol, a single antigen mismatch at the HLA A, B, C, with or without additional single allele level mismatch may participate in this protocol for voluntary unrelated donors (blood or marrow) DONOR: Donor must be healthy and have non-reactive test results for all infectious disease assays as required by state and federal regulations; donors who screen seropositive for hepatitis an/or syphilis must be cleared by infectious disease consultation DONOR: Donor must have no uncontrolled cardiopulmonary, renal, endocrine, hepatic or psychiatric disease to render donation unsafe DONOR: The donor (or parent in minor) must give informed consent for peripheral blood stem cell collection or bone marrow collection DONOR: Syngeneic donors are not eligible DONOR: Donors who have poor peripheral venous access, may require central venous line placement for stem cell apheresis

Exclusion Criteria:

* Uncontrolled central nervous system (CNS) disease (for hematologic malignancies)
* Karnofsky (adult) or Lansky (for =< 16 years) performance status < 50%
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 40% predicted, corrected for hemoglobin and/or alveolar ventilation
* Left ventricular ejection fraction < 40% - Bilirubin >= 3 X upper limit of normal
* Liver alkaline phosphatase >= 3 x upper limit of normal
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvate transaminase (SGPT) >= 3 x upper limit of normal
* Child's class B and C liver failure
* Calculated creatinine clearance < 40 cc/min by the modified Cockroft-Gault formula for adults or the Schwartz formula for pediatrics
* Patients who have received maximally allowed doses (given in 2 Gy fractionations, or equivalent) of previous radiation therapy to various organs as follows: * Mediastinum: adult -40, pediatric (=<18 yrs) - 21 * Heart: adult 36, pediatric - 26 * Whole lung(s): adult - 12, pediatric - 10 * Small bowel: adult - 46, pediatric - 40 * Kidneys: adult - 12, pediatric - 10 * Whole liver: adult - 20, pediatric - 20 * Spinal cord: adult - 36, pediatric - 36 * Whole Brain: adult 30, pediatric - 30
* Patients who previously have received a higher than allowed dose of radiation to a small lung, liver, and brain volume, will be evaluated by the radiation oncologist to determine if the patient is eligible for study
* Uncontrolled diabetes mellitus, cardiovascular disease, active serious infection or other condition which, in the opinion of treating physician, would make this protocol unreasonably hazardous for the patient
* Human immunodeficiency virus (HIV) positive
* Patients who in the opinion of the treating physician are unlikely to comply with the restrictions of allogeneic stem cell transplantation based on formal psychosocial screening
* Female of childbearing potential with a positive pregnancy test

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-02-28 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Chen, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Started | 94
Completed | 94
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Number analyzed (Participants) | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 66
  >=65 years | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 93
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Transplant Related Mortality (TRM)
Description: Day 100 transplant related mortality (TRM). An exact 95% confidence interval will be provided.
Time Frame: In the first 100 days from day 0 of transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Number analyzed (Participants) | 94
percentage of participants | 8.5 [4.0 to 15.3]

2. Secondary Outcome: Clinical Response
Description: Patients will be followed according to response criteria as referenced in BMT SOP "Standards of Therapy" last updated 2008. Clinical Response = CR + PR.
  Complete Response Requires all of the following:
  * Serum and urine negative for monoclonal proteins by immunofixation
  * Normal free light chain ratio
  * Plasma cells in marrow < 5%
  Partial Response (PR) Requires any of the following:
  - ≥ 50% reduction in current serum monoclonal protein levels > 0.5 g/dL or urine light chain levels > 100 mg/day with a visible peak or free light chain levels > 10mg/dL
  Progressive Disease (PD) Requires any of the following:
  * If progressing from CR, any detectable monoclonal protein or abnormal free light chain ratio (light chain must double)
  * If progressive from PR or SD, ≥ 50% increase in the serum M protein to > 0.5 g/dL,or ≥ 50% increase in urine M protein to > 200mg/day with visible peak present.
  * Free light chain increase of ≥ 50% to
Time Frame: In the first 100 days from day 0 of transplant
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Number analyzed (Participants) | 94
percentage of participants | 45 [34 to 55]

3. Secondary Outcome: Progression Free Survival (PFS) at One Year
Description: Assessed using Kaplan Meier and Proportional Hazards
Time Frame: day of transplant until progression up to 5 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Number analyzed (Participants) | 94
percentage of participants | 85 [76 to 91]

4. Secondary Outcome: Median Time to Neutrophil Engraftment
Description: Median time to recovery of absolute neutrophil count >=500/uL for 3 consecutive days. Summarized using standard descriptive statistics along with corresponding 95% confidence intervals.
Time Frame: Day 100
Population: All treated and eligible patients
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Number analyzed (Participants) | 94
days | 17 [6 to 64]

ADVERSE EVENTS:
Arm/Group | Treatment (Reduced Intensity Allogeneic PBSCT)
Serious Adverse Events (participants affected / at risk) | 17/94
Other Adverse Events (participants affected / at risk) | 1/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Reduced Intensity Allogeneic PBSCT) (N=94)
Myocardial infarction (Cardiac disorders) | 1 (4)
Multi-organ failure (General disorders) | 1 (8)
Pyrexia (General disorders) | 2 (22)
Acute graft versus host disease in intestine (Immune system disorders) | 2 (18)
Graft versus host disease (Immune system disorders) | 3 (13)
Infection (Infections and infestations) | 1 (5)
Pneumonia (Infections and infestations) | 1 (8)
Blood culture positive (Investigations) | 1 (4)
Gram stain positive (Investigations) | 1 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (4)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Hospitalisation (Surgical and medical procedures) | 1 (4)
Hypotension (Vascular disorders) | 1 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Reduced Intensity Allogeneic PBSCT) (N=94)
Acute graft versus host disease in intestine (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-10-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT01529827/Prot_SAP_000.pdf
  • Informed Consent Form (2014-09-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT01529827/ICF_001.pdf